CLINICAL TRIAL: NCT01947790
Title: Pioglitazone Regress Left Ventricular Mass in Type 2 Diabetes With Ischeamia Heart Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Pioglitazone regress the left ventricular mass in normotensive type 2 diabetic patients with ischeamia heart disease, Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013Wze051
Record Dates: First submitted 2013-09-02; First posted 2013-09-20 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: LVM; Type 2 Diabetic Patients With IHD; Endothelial Function
Keywords: Type 2 diabetes; left ventricular mass; pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone group (Experimental): Pioglitazone 15 mg/day will be given in this group for 9 months
  Interventions: Drug: pioglitazone group
- Metformin group (Active Comparator): Metformin 0.85 twice daily will be given in this group for 9 months as control.
  Interventions: Drug: Metformin group

INTERVENTIONS:
Drug: pioglitazone group
  Arms: Pioglitazone group
Drug: Metformin group
  Arms: Metformin group

SUMMARY:
Cardiovascular complications account for the highest mortality in type 2 diabetic patients, mainly due to ischeamia heart disease (IHD). Most of the attention in treating IHD in type 2 diabetes is understandably directed toward treating coronary artery conditions. However there are other treatable culprits in these patients.

Left ventricular hypertrophy (LVH) is widespread in type 2 diabetic patients with IHD, even in the absence of hypertension. It is a strong predictor of cardiovascular events and all-cause mortality. In one study, the presence of LVH was a stronger predictor of mortality than either multivessel coronary disease or impaired left ventricular function. Regression of LVH has been associated with an improved prognosis, independent of change in blood pressure (BP). Therefore, cardiovascular events and mortality in type 2 diabetes with IHD might will be reduced if we can find novel therapies to regress LVH.

Pioglitazone can improve atherosclerosis. Therefore, we hypothesied that pioglitazone can regress the left ventricular mass (LVM) in type 2 diabetes with IHD.Therefore, in this study, we will treat patients with pioglitazone, and we will also metformin as control.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* aged 40～75 years old
* with IHD

Exclusion Criteria:

* heart failure
* renal failure
* hypertension (>130/80 mmHg)
* hemoglobin A1c 9%

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The changes of LVM | The LVM will be measured at baseline, 6 momth and 9 month

SECONDARY OUTCOMES:
The changes of endothelial function | The endothelial function will be measured at baseline, 6 month and 9 month

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Wuhan, Hubei
  - Xiang Guangda, Wuhan, Hubei